CLINICAL TRIAL: NCT06781463
Title: Creation of a Prospective Data Collecting Registry for Genicular Artery Embolization for Arthritis (GAE)
Brief Title: Creation of a Prospective Data Collecting Registry for Genicular Artery Embolization for Arthritis
Acronym: GAE
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB22-1164
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis; Knee Osteoarthritis (Knee OA); Knee Osteoarthritis (OA)
Keywords: knee pain; knee replacement alternative; knee arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry: Since this is a registry all enrolled patients are part of one group and will be followed for one year from the respective date of procedure.
  Interventions: Other: Registry (N/A)

INTERVENTIONS:
Other: Registry (N/A) — This study is a registry, thus no research intervention is being directly tested.

SUMMARY:
The goal of this study is to create a prospective registry (<100 patients) to show the effectiveness of the genicular artery embolization procedure overtime in reducing bilateral or unilateral osteoarthritic knee pain as measured by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a pervasive and debilitating disease, affecting over 15 million people in the US alone. Symptoms include pain, stiffness, and ultimately loss of joint function. Medical therapies are the mainstay of treatment as surgical joint replacement is typically reserved for advanced disease. Only half of patients treated by medical management with disease not severe enough to warrant surgery experience adequate pain relief, resulting in an estimated population of 3.6 million Americans who are left suffering. Genicular artery embolization (GAE) is a novel, minimally invasive treatment that uses radiologic techniques to catheterize pathologically hyperemic genicular arteries using live X-ray guidance with subsequent occlusion of these vessels using injected microspheres. GAE is performed to inhibit or blunt synovial inflammation thought to be a primary phenotype of KOA. Multiple small sized cohort studies have shown to significantly reduce pain associated with KOA. This procedure has been performed in the University of Chicago Medical Center and showed its effectiveness and safety. In this study, the investigators plan to establish a prospective database of patients undergoing GAE for KOA in order to further characterize its effectiveness with a longer follow-up and larger sample size. The investigators also hope to establish Magnetic Resonance Imaging (MRI) as an objective imaging biomarker for positive remodeling of the knee that occurs after GAE due to decreased synovitis. If the results of this study are positive, the investigators plan to conduct a definitive sham-controlled study to justify the use of GAE in medically refractory KOA and help provide a treatment option to the millions of people with this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >=18
* Bilateral or unilateral knee pain attributed to knee osteoarthritis (KOA). For bilateral KOA patients, the more severe knee will be permitted inclusion to the registry
* Grade 1-3 Osteoarthritis as diagnosed on standing weight-bearing knee radiographs per the Kellen-Lawrence Grading scale
* Knee pain >6 months refractory to conservative medical management (Nonsteroidal anti-inflammatory drugs, acetaminophen, etc.)
* Not eligible for surgical knee replacement or patient's personal preference to undergo Genicular Artery Embolization (GAE) for reasons such as minimally invasiveness of GAE

Exclusion Criteria:

* Active malignancy
* Active infection of the affected knee
* Platelets <50,000/uL, INR >2.0 (unless on anticoagulation that can be reversed or performing radial/pedal access without reversal)
* Corticosteroid injection of the affected knee within 3 months of enrollment
* Rheumatoid arthritis or other seronegative arthropathy
* Previous surgery (excluding arthroscopy) of the affected knee
* Grade 4 per Kellgren-Lawrence Grading Scale of the affected knee
* Pregnancy or expected pregnancy
* Glomerular Filtration Rate (GFR) <30
* Anaphylactic reaction to iodinated contrast
* Moderate to severe pain in other lower limb joints
* Body weight >400 lbs. (prohibiting safe angiography)
* Peripheral arterial disease of the treated extremity (Rutherford Grade 2 or greater)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with medically refractory knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 1 year of enrollment/patient
  The investigators will describe differences in pain response with Genicular Artery Embolization (GAE) compared to a sham procedure when treating medically refractory mild to moderate Knee Osteoarthritis (KOA) at 12 months as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale score. A higher score index a higher pain level while a lower score indicates lower pain levels. The score range is 0 to 100.

SECONDARY OUTCOMES:
Incidence of Genicular Artery Embolization Emergent Adverse Events | 1 year of enrollment/patient
  The investigators will assess GAE-related adverse events to better understand its net benefit. Angiography with embolization is an invasive procedure with knowns risks that include bleeding (i.e. hematoma, arterial perforation), infection, and non-target embolization.35 Outcomes will be recorded as intra-procedure events along with assessments at 3, 6, 9, and 12 months post procedure. Complications will be recorded per the Society of Interventional Radiology Quality Improvement Standards for Percutaneous Transcatheter Embolization.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Duchossois Center for Advanced Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
All IPD is de-identified when entered into the EDC. Results will not share IPD or PHI, rather the trends and calculations that are concluded based on data collected in the EDC.

REFERENCES:
- [Background] Berenbaum F. Osteoarthritis as an inflammatory disease (osteoarthritis is not osteoarthrosis!). Osteoarthritis Cartilage. 2013 Jan;21(1):16-21. doi: 10.1016/j.joca.2012.11.012. Epub 2012 Nov 27. PMID 23194896
- [Background] London NJ, Miller LE, Block JE. Clinical and economic consequences of the treatment gap in knee osteoarthritis management. Med Hypotheses. 2011 Jun;76(6):887-92. doi: 10.1016/j.mehy.2011.02.044. Epub 2011 Mar 25. PMID 21440373
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Litwic A, Edwards MH, Dennison EM, Cooper C. Epidemiology and burden of osteoarthritis. Br Med Bull. 2013;105:185-99. doi: 10.1093/bmb/lds038. Epub 2013 Jan 20. PMID 23337796
- See also: UChicago Knee Osteoarthritis WebPage — https://www.uchicagomedicine.org/conditions-services/orthopaedics/knee-care/genicular-artery-embolization